CLINICAL TRIAL: NCT01900288
Title: Mobile Technologies Assisting Patients & Family Caregivers in Healthy Living
Brief Title: Home Parenteral Nutrition (HPN) Families' Mobile Distance Connections to Care Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13337; R01EB015911 (NIH)
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Short Bowel Syndrome; Malabsorption; Malnutrition
Keywords: short bowel disorder; short bowel syndrome; home parenteral nutrition; HPN; total parenteral nutrition; TPN; telehealth; telemedicine
MeSH Terms: conditions — Short Bowel Syndrome; Malabsorption Syndromes; Malnutrition; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPN Group Clinic Appointments (Group 1) (Experimental): A mobile device (iPad mini) is loaned to Group 1 subjects providing a connection to HPN Internet information for the 6 to 12 months of the study. Two scheduled times during the study period, visual connections to geographically distant professionals and peers over the iPad mini (HPN Group Clinic Appointment) will be held for approximately 1 ½ to 2 hours each time (called Healthy Living Connections).
  On the iPad mini screen during the HPN Group Clinic Appointments, subjects will be able to see professionals and peers all at the same time and they will be able to see them in their home. This group will also receive electronic prompts about healthy activities.
  Interventions: Behavioral: HPN Group Clinic Appointments using Mobile Devices (experimental)
- Mobile Device Access (Group 2) (Placebo Comparator): A mobile device (iPad mini) is loaned to Group 2 subjects providing a connection to Internet information for the 6 to12 months of the study. At the end of the study period, Group 2 subjects will have 1 scheduled time during the study to connect to professionals and peers over the iPad mini for approximately 1 ½ to 2 hours (called Healthy Living Connections) before the study concludes.
  On the iPad mini screen during the placebo control group clinics, subjects will be able to see professionals and peers all at the same time and they will be able to see them in their home. This group will also receive one electronic prompt about healthy activities as a comparison control to the intervention group.
  Interventions: Behavioral: Mobile Device Access (placebo)

INTERVENTIONS:
Behavioral: HPN Group Clinic Appointments using Mobile Devices (experimental) — Visual meetings with geographically distant professionals and peers using a mobile device (iPad mini).
  Other Names: Healthy Living Connections
  Arms: HPN Group Clinic Appointments (Group 1)
Behavioral: Mobile Device Access (placebo) — Use of iPad mini unrelated to the intervention until last contact with one connection to professionals for comparison.
  Other Names: Placebo use of a mobile device
  Arms: Mobile Device Access (Group 2)

SUMMARY:
The purpose of this study is to test Mobile Technologies in Assisting Patients & Family Caregivers in Healthy Living and complex home care by connecting to information and professionals from a distance.

DETAILED DESCRIPTION:
HPN (Home Parenteral Nutrition) families with TPN (Total Parenteral Nutrition) users are typically geographically distant from one another (peers) as well as professional providers. Real-time mobile access to health related information, peer and professional support will be tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* 13 years or older total parenteral nutrition (TPN) patients/users and family members/caregivers (defined as those individuals involved in daily home HPN care)
* TPN users (also called HPN users) must be receiving intravenous nutrition for a non-malignant short bowel disorder
* Read, write, speak English and provide informed consent
* Be able to participate in group clinic visits

Exclusion Criteria:

* enteral nutrition dependency only
* less than 13 years of age
* 13 through 17 years of age without parental consent
* currently enrolled in an intervention study or HPN management program
* severe cognitive impairment
* disability disorders (e.g. blindness which cannot be accommodated for active participation in the group clinics

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2016-12-23 (Actual)

PRIMARY OUTCOMES:
Engagement in Healthy Living Activities | 4 Months
  Change from Baseline to 4 Months of the logged frequency of healthy living activities with a 10-item Likert scale.
Health Satisfaction SF-12 | 4 Months
  Change from Baseline to 4 Months of the Health Survey SF-12v2 7-item Likert scale rating.
Quality of Life | 4 Months
  Change from Baseline to 4 Months of the 3-item Likert scale rating using the Cantril Ladder.
Access to Health Care | 4 Months
  Change from Baseline to 4 Months of the 6-item Likert scale instrument rating.
Engagement in Healthy Living Activities | 8 Months
  Change from Baseline to 8 Months of the logged frequency of healthy living activities with a 10-item Likert scale.
Health Satisfaction SF-12 | 8 Months
  Change from Baseline to 8 Months of the Health Survey SF-12v2 7-item Likert scale rating.
Quality of Life | 8 Months
  Change from Baseline to 8 Months of the 3-item Likert scale rating using the Cantril Ladder.
Access to Health Care | 8 months
  Change from Baseline to 8 Months Change of the 6-item Likert scale instrument rating.

SECONDARY OUTCOMES:
Preparedness to Manage Home-Care | 4 Months
  Change from Baseline to 4 Months of the caregiver strain rating with and 8-item Likert scale.
Caregiving Burden | 4 Months
  Change from Baseline to 4 Months of the rating from the Oberst Caregiving Burden Scale 15-item Likert scale.
Preparedness to Manage Home-Care | 8 Months
  Change from Baseline to 8 Months Change from Baseline to 4 Months of the caregiver strain rating with and 8-item Likert scale.
Caregiving Burden | 8 Months
  Change from Baseline to 8 Months Change from Baseline to 4 Months of the rating from the Oberst Caregiving Burden Scale 15-item Likert scale.
Virtual Nurse Caring | 8 months
  At 8 months, using the Virtual Nurse Caring 20-item Likert scale instrument, caregiver's rating of perception of nurse care and needs met via mobile device is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Smith, RN PhD FAAN, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States